CLINICAL TRIAL: NCT05808881
Title: Clinical Outcomes From Injectable Nalmefene in the Emergency Department (COINED)
Brief Title: Clinical Outcomes From Nalmefene
Acronym: COINED
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to changes in research objectives and methodological approach.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAL4001
Record Dates: First submitted 2023-03-15; First posted 2023-04-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose | interventions — nalmefene; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nalmefene (Experimental): Nalmefene hydrochloride (HCl) injection
  Interventions: Drug: Nalmefene Hydrochloride Injection
- Naloxone (Active Comparator): Naloxone hydrochloride (HCl) injection
  Interventions: Drug: Naloxone Hydrochloride Injection

INTERVENTIONS:
Drug: Nalmefene Hydrochloride Injection — for intravenous/intramuscular/subcutaneous (IV/IM/SC) administration
  Arms: Nalmefene
Drug: Naloxone Hydrochloride Injection — for intravenous/intramuscular/subcutaneous (IV/IM/SC) administration
  Other Names: Narcan
  Arms: Naloxone

SUMMARY:
The purpose of this study is to assess the effectiveness of nalmefene relative to naloxone for the reversal of opioid intoxication in emergency department (ED) settings.

ELIGIBILITY:
Inclusion Criteria:

1. Presumed or known opioid overdose in community settings.
2. Experiencing clinically significant respiratory depression based on appropriate medical judgement.
3. Patient airway is open and unobstructed at the time of enrollment. (Utilization of oral pharyngeal or nasal pharyngeal airway is allowed.)
4. Pre-hospital naloxone administration is allowed.

Exclusion Criteria:

1. Patient age known or estimated to be less than 18 years.
2. Patient has one or more additional documented acute medical, traumatic, toxicologic, or psychiatric conditions that would extend length of treatment or adversely alter the clinical outcome.
3. Cardiac arrest, secondary to opioid intoxication.
4. Arrested, jailed, or imprisoned patients.
5. Inappropriate for the study per judgement of research team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Reversal of Respiratory Depression | Up to 3 hours
  Normalization of the end tidal carbon dioxide value (if measured) to between 35 and 45 mmHg
  and/or
  ≥5 breaths per minute increase in respiratory rate from baseline (pre-dose) measurement, with rate of at least 12 breaths per minute.

SECONDARY OUTCOMES:
Time to Reversal from administration of opioid antagonist | Up to 3 hours
Recurrence of Respiratory Depression | Up to 3 hours
  Increased end tidal carbon dioxide value (if measured) above 45 mmHg when previously within the normal range
  and/or
  ≥5 breaths per minute decrease in respiratory rate from maximum post-reversal measurement, with a rate of at most 12 breaths per minute.
ED Disposition | Up to 3 hours
  One of the following will apply:
  * ED Discharge
  * Hospital Admission
  * ICU Admission
  * Left against medical advice
  * Transfer to another facility
  * Death.
Drug Dosing | Up to 3 hours
  1. Dose administered for each opioid antagonist given to patients during their ED encounter -
     * Individual dose amount and frequency
     * Cumulative dose
  2. Any pre-hospital naloxone given prior to ED arrival -
     * Dose amount, route
Richmond-Agitation Sedation Scale (RASS) Score | Up to 3 hours
  This is a single-item instrument used to quickly assess the degree of patient alertness and agitation in emergency and critical care settings. It is an observational assessment conducted by healthcare providers, and it can be completed in seconds. The scale uses integers from -5 to +4, each with its own clear anchor. A score of 0 means that the patient is alert and calm. Negative integers indicate diminished responsiveness and consciousness, with -1 indicating that a patient will open their eyes or make eye contact for 10 or more seconds when awakened by voice, and -5 meaning that the patient is unarousable by voice or physical stimulation. Positive integers indicate an increased level of arousal or agitation. The positive end of the scale spans from +1 (anxious, apprehensive, but not aggressive) to +4 (combative, violent, danger to staff).
Clinical Opioid Withdrawal Scale (COWS) Score | Up to 3 hours
  This is an observational assessment performed by a clinician to diagnose and assess the severity of opioid withdrawal symptoms. Eleven different opioid withdrawal symptoms are included in the COWS. The clinician will score the presence and severity of each symptom, with 0 indicating that the symptom is absent and more severe symptoms warranting a higher score. Individual symptom scores are then added to determine the overall severity of the patient's withdrawal. Total scores range from 5 to 48 where 5 - 12 = mild; 13 - 24 = moderate; 25 - 36 moderately severe; and greater than 36 = severe withdrawal.
Oxygen saturation level | Up to 3 hours
  Pulse oximetry monitoring will be used to assess the patient's oxygen saturation level (SpO2), expressed as a percentage from 0 to 100.
Length of time during ED encounter | Up to 3 hours
  Defined as the difference between time at Triage to time at ED Disposition

IPD SHARING:
Plan to Share IPD: No